CLINICAL TRIAL: NCT01538758
Title: Treatment of Calcifying Tendinitis of the Shoulder: Ultrasound Guided Needling With Subacromial Corticosteroid Injection Versus Ultrasound Guided Subacromial Corticosteroid Injection Only, a Randomized Controlled Trial.
Brief Title: Ultrasound Guided Needling Versus Ultrasound Guided Corticosteroid Injection Alone, a Randomized Controlled Trial.
Acronym: BARB-01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medisch Spectrum Twente (Other)
Responsible Party: Principal Investigator, Eva Genbrugge, Principal investigator, Medisch Spectrum Twente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P12-03
Record Dates: First submitted 2011-11-30; First posted 2012-02-24 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Calcific Tendinitis
Keywords: calcifying tendinitis; rotator cuff
MeSH Terms: interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Us guided needling (Active Comparator): Us guided needling is a therapeutical technique treating calcifying tendinitis of the shoulder. Calcifications in the rotator cuff tendon are visualised with ultrasound. Under ultrasound guidance a 20 gauge needle is inserted in the calcification. Lidocaine 1% in a 1cc syringe is injected in the calcification and aspirated. The calcification is flushed until the fluid is clear. Sometimes it is not possible to flush the calcification. In this case the calcification will be fragmented.
  After flushing or fragmentation of the calcification, 20 mg triamcinolone with 1cc lidocaine 1% will be injected in de subacromial bursa under us guidance.
  Interventions: Other: Us guided needling
- corticosteroid injection (Active Comparator): Us guided subacromial bursa injection with 20 mg triamcinolone with 1cc lidocaine 1%.
  Interventions: Other: corticosteroid injection

INTERVENTIONS:
Other: Us guided needling — Us guided needling is a therapeutical technique treating calcifying tendinitis of the shoulder. Calcifications in the rotator cuff tendon are visualised with ultrasound. Under ultrasound guidance a 20 gauge needle is inserted in the calcification. Lidocaine 1% in a 1cc syringe is injected in the calcification and aspirated. The calcification is flushed until the fluid is clear. Sometimes it is not possible to flush the calcification. In this case the calcification will be fragmented.
  After flushing or fragmentation of the calcification, 20 mg triamcinolone with 1cc lidocaine 1% will be injected in de subacromial bursa under us guidance.
  Other Names: Barbotage
  Arms: Us guided needling
Other: corticosteroid injection — Us guided subacromial bursa injection with 20 mg triamcinolone with 1cc lidocaine 1%.
  Arms: corticosteroid injection

SUMMARY:
Ultrasound guided needling is becoming an accepted treatment for patients with shoulder pain due to calcifying tendinitis. However, evidence for this treatment is lacking. The investigators expect that patients treated with us guided needling with corticosteroid injection compared with patients treated with only corticosteroid injections in the subacromial bursa have better clinical outcome after one year follow-up.

DETAILED DESCRIPTION:
Calcifying tendinitis of the shoulder is a common cause of shoulder pain with an incidence ranging from 2.7 % to 6.8 %. This disease of the rotator cuff tendons is characterised by calcifications in the tendons, most commonly in the supraspinatus tendon up to 82%. The aetiology remains unclear.

Calcifying tendinitis is regarded as a self-healing condition with usually spontaneous resolution of the calcifications. But some patients have chronic or recurrent pain and disability of the shoulder which requires treatment. The treatment should be minimally invasive and effective in short and long term. Symptomatic treatment is indicated first using non-steroidal anti-inflammatory drugs, therapeutic exercise and non ultrasound guided subacromial corticosteroids injection.

The role of corticosteroid injections is unknown due to the lack of good studies. Family doctors and orthopaedic surgeons inject corticosteroids in the shoulder without the guidance of ultrasound; with this method accurate needle placement in the subacromial bursa is not possible. When this treatment fails other therapeutical methods can be used. Ultrasound guided needling is a percutaneous technique of fragmentation or extraction of calcifications in the rotator cuff tendon.

Literature shows favourable results but only a few randomized controlled trials were executed. Randomised controlled trials are needed to give more insight in the effectiveness of us guided needling. Comparing two groups of patients treated with us guided corticosteroid injection and one group combined with us guided needling can provide information of the usefulness of us guided needling.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder pain without improvement after 3 months despite conservative treatment
* Calcification on x-ray (Gartner type I of II) and ultrasound in the supraspinatus tendon less than 6 weeks before the treatment
* All patients are first seen and included by the orthopaedic surgeon

Exclusion Criteria:

* Previous operation of the shoulder
* Previous ultrasound guided needling of the shoulder
* Frozen shoulder
* Last corticosteroid injection less than 3 months ago
* Comorbidities of the painful shoulder on x-ray or ultrasound ( ruptured tendon, fracture, bursitis,...)
* No informed consent
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
VAS score on long term | 1 year
Constant score on long term | 1 year
  The constant score is a validated scale, measuring the shoulder function. It is a objective measurement independent of the shoulder pain.

SECONDARY OUTCOMES:
Constant score | baseline,6 weeks, 3 months and 6 months
  To have a more insight over time the constant score will be measured at baseline, 6 weeks, 3 months and 6 months
VAS score | Baseline, 2 weeks, 6 weeks, 3 months and 6 months
  To have a more insight over time the VAS score will be measured at baseline, 6 weeks, 3 months and 6 months.
  In practice patients seem to have a maximum pain shortly after the us guided needling. To measure this a VAS score will be taken after two weeks.
DASH score | baseline, 6 weeks, 3 months, 6 months and 1 year.
  This score measures the disability of the shoulder in daily life, work, sports and hobby over time.
Gärtner score of the shoulder calcifications on x-ray | at baseline, directly post-interventional, at 6 weeks and one year.
Scoring system presented by Chiou et all. of the calcifications of the supraspinatus tendon on ultrasound | at baseline, directly post-interventional, at 6 weeks and one year.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Genbrugge, MD, Principal Investigator — MST
Locations (1):
- Medisch Spectrum Twente, Enschede, Netherlands